CLINICAL TRIAL: NCT05891457
Title: Changes in the Nerve Electro Physiologic Properties Before and After Correction of Malnutrition in Under-5 Children
Brief Title: Changes in Nerve Electro Physiologic Properties in Children Before and After Correction of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-21013
Record Dates: First submitted 2023-05-22; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Stunting; Severe Acute Malnutrition; Wasting
Keywords: Malnutrition; Nerve Conduction
MeSH Terms: conditions — Growth Disorders; Severe Acute Malnutrition; Cachexia; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malnourished children (Experimental): * Severe Stunting (length/height-for-age Z-scores <-3SD)
  * Severe Acute Malnutrition (weight-for-length/height Z-scores <-3SD, and/or mid-upper-arm circumference <11.5 cm, with or without nutritional edema)
  * Wasting (weight-for-length/height Z-scores<-3SD)
  Interventions: Combination Product: Nutritional Intervention

INTERVENTIONS:
Combination Product: Nutritional Intervention — * Severe acute malnourished children were provided with appropriate nutritional therapy/treatment that include supplementation of a high-calorie diet; i.e., F-100 milk and khichuri-halwa for nutritional rehabilitation.
  * Egg milk and micronutrient supplementation for recovery from severe stunting following standard guidelines for facility based management and recently conducted community based nutrition intervention studies.
  * Wasted children were treated with suitable local nutritional management (NM), such as infant and young child feeding practices (IYCF), providing MNP and nutrition education.

SUMMARY:
The goal of this clinical trail study is to measure neurophysiologic parameters to assess the effect of malnutrition on the peripheral nervous system and their response to treatment in three categories (SAM, severe wasting, and severe stunting) of childhood malnutrition. 83 under-5 children from three categories of undernourished groups- severe stunting (n=30), Severe acute malnourished (n=22), wasting (n=31), and 45 age-matched healthy children from urban/peri-urban areas were enrolled.

SAm were provided with appropriate nutritional therapy/treatment that include supplementation of a high-calorie diet; i.e., F-100 milk and khichuri-halwa for nutritional rehabilitation. Egg milk and micronutrient supplementation were for recovery from severe stunting. Wasted children were treated with suitable local nutritional management (NM), such as infant and young child feeding practices (IYCF), providing MNP and nutrition education. Wasted children with medical complications were treated with specialized therapeutic milk (F-75) and those without medical complications were treated with a suitable local Nutritional Management (NM) & routine medicines to treat simple medical conditions at community nutrition center (CNC) with weekly follow up. At day 60 of intervention, children were again brought to icddr,b for a nerve conduction test.

DETAILED DESCRIPTION:
The purpose of this study is to measure neurophysiologic parameters to assess the effect of malnutrition on peripheral nervous system and their response to treatment in three categories (SAM, severe wasting and severe stunting) of childhood malnutrition. The electrophysiological properties of peripheral nerves in malnourished under-5 children before and after correction of severe malnutrition were assed.

This is an exploratory study conducted in icddr,b, Dhaka, Bangladesh. 83 under-5 children from three categories of undernourished groups- severe stunting (length-for-age Z-scores <-3), SAM (weight-for-length Z-scores <-3, and/or mid-upper-arm circumference <11.5 cm, with or without nutritional edema) and wasting (weight-for-length Z-scores (WLZ) <-2) were enrolled. A total of 45 age-matched healthy children selected as controls. Participants were identified from urban/peri-urban areas of Dhaka city. After enrolment, participants were brought to icddr,b Dhaka Hospital and data on socio-economic status, weaning practice, morbidity, and dietary intake were collected. Nerve electro physiologic parameters assessed by motor (median, ulnar, fibular and tibial) and sensory (median, ulnar and sural) nerve conduction studies (NCS) on enrollment.

SAM were treated with appropriate nutritional therapy/treatment that included supplementation of high calorie diet; i.e., F-100 milk and khichuri-halwa for nutritional rehabilitation. Egg-milk and micronutrient supplementation were provided for 2 months for recovery from severe stunting (following standard guidelines for facility based management and recently conducted community based nutrition intervention studies). As per national guidelines, children suffering from severe wasting with medical complications were treated with specialized therapeutic milks (F-75) and those without medical complications treated with a suitable local Nutritional Management (NM) & routine medicines to treat simple medical conditions at community nutrition center (CNC) with weekly follow up. Children were monitored in the community for 2 months. Monthly anthropometry had been done. On day 60 or 2 months of intervention, children with weight-for-length/height Z-scores ≥-1 and MUAC >115 mm were again brought to icddr, b for nerve conduction test.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will give informed written consent
* Children aged between 6 months to 5 years of age
* Children whose length/height-for-age <-3 (Stunted), weight-for-length/height <-2 (Wasted), and weight-for-length/height z scores <-3 and/or mid upper arm circumference <11.5 cm, with or without nutritional edema
* Children whose length/height-for-age, weight-for-length/height, and weight-for-length/height z score will be ≥1

Exclusion Criteria:

* Participants with congenital anomalies, twins and multiple pregnancies

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Compound muscle action potential (CMAP) amplitude | 60 days
  Motor nerve compound muscle action potential (CMAP) amplitude is measured from baseline to peak amplitude for all the stimulation sites and expressed in millivolts (mV)
Motor nerve conduction velocity | 60 Days
  Motor nerve conduction velocity is measured by the distance between the distal and proximal stimulation sites, divided by the difference in latency, and expressed in meters per second (m/s)
Motor nerve corrected distal latency | 60 Days
  Motor nerve corrected distal latency is measured from the onset (or rise of the negative deflection) of the compound muscle action potential and expressed in milliseconds (ms)
Sensory nerve action potential (SNAP) amplitude | 60 Days
  Sensory nerve action potential (SNAP) amplitude is measured from baseline-to-peak amplitude at the distal stimulation site and expressed in microvolts (μV)
Sensory nerve conduction velocity | 60 Days
  Sensory nerve conduction velocity is measured by the distance between the distal and proximal stimulation sites, divided by the difference in latency, and expressed in meters per second (m/s)
Sensory nerve corrected distal latency | 60 Days
  Sensory nerve corrected distal latency is measured from the onset (or rise of the negative deflection) of the compound muscle action potential and expressed in milliseconds (ms).

SECONDARY OUTCOMES:
Changes in weight | 60 Days
  Changes in weight measured in kg
Changes in height | 60 Days
  Changes in height measured in cm
Changes in Mid Upper Arm Circumference (MUAC) for SAM | 60 Days
  Changes in Mid Upper Arm Circumference (MUAC) measured in mm or cm
Changes in weight-for-height Z score for SAM | 60 Days
  Changes in weight-for-height Z score measured in points
Changes in weight-for-height Z score for Wasted | 60 Days
  Changes in weight-for-height Z score measured in points
Changes in height-for-age Z score for Stunted | 60 Days
  Changes in height-for-age Z score measured in points

CONTACTS AND LOCATIONS:
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naila NN, Hossain MS, Alam A, Das S, Karmakar G, Mahfuz M, Ahmed T, Islam B. Nutritional Intervention Improves Nerve Conduction in Malnourished Children Under 5 Years of Age. Acta Paediatr. 2025 Nov;114(11):2864-2873. doi: 10.1111/apa.70179. Epub 2025 Jun 18. PMID 40530465